CLINICAL TRIAL: NCT00739271
Title: Early Enteral Feeding After Intestinal Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Responsible Party: Dr. Rajeev Kapoor, CMC Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RK2
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Intestinal Anastomosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study arm (Active Comparator): Early enteral feed 48 hours after abdominal surgery
  Interventions: Other: Early feeding
- Control arm (Active Comparator): Traditional treatment where patient is kept on a nasogastric drainage for a few days after abdominal surgery, wait for bowel sounds to appear and then start enteral feeds.
  Interventions: Other: late feeding after bowel sounds return

INTERVENTIONS:
Other: Early feeding
  Arms: Study arm
Other: late feeding after bowel sounds return — Traditional method
  Arms: Control arm

SUMMARY:
The concept of starting the patient on early enteral nutrition has been a topic of much interest and research in the past decade. It is gaining widespread acceptance worldwide as more and more studies are being conducted proving early enteral nutrition to be more physiological, to prevent morphologic and functional trauma related alterations of the gut and to modulate immune and inflammatory responses, and as being less expensive than total parenteral nutrition. Early enteral nutrition is a major component of the recently introduced post operative rehabilitative regimens.

Early feeding has been shown to reduce the risk of any specific infection, mean length of hospital stay, anastomotic dehiscence, wound infection, pneumonia, intra abdominal abscesses. It leads to lower weight loss and early positive nitrogen balance. Hence, overall early enteral nutrition leads to reduced post operative morbidity and better patient outcome.

The objective of this study was to study and compare the effects of early enteral feeding with those of conventional management in patients undergoing intestinal anastomosis; the end points being return of bowel activity, incidence of septic complications, length of hospital stay, weight loss and post operative morbidity.

DETAILED DESCRIPTION:
Pre operatively, common parameters observed in both study and control groups were:

* Name
* Age
* Sex
* Date of admission
* Weight
* Indication of surgery
* Pre operative features of sepsis (whether present or not) which included temperature, pulse rate& total leukocyte count.

Post operatively, the patients in the study group were kept nil per orally for the first forty eight hours. The nasogastric tube was removed on the first post operative day invariably.

After forty eight hours of surgery, subjects were started on sips of clear liquids orally; the amount was gradually increased as tolerated by the patient. The diet was stepped up to soft diet and to regular diet. A record was made of abdominal discomfort, pain or distension if experienced by the subject during feeding.

Record was made of the following:

* Site of anastomosis
* Type of anastomosis ( sutured / stapled )
* Time of removal of nasogastric tube
* Time of passage of flatus / stools post operatively
* Time of appearance of bowel sounds
* Features of sepsis which included temperature, pulse rate & total leukocyte count
* Presence of wound infection
* Weight on the fifth day of surgery, at the time of discharge
* Date of discharge
* Length of hospital stay

Patients in the control group were kept on maintenance intravenous fluids containing dextrose and saline. Nasogastric tube was removed and feeds were started orally as decided by the operating surgeon depending on the clinical condition of the patient and presence of bowel activity. Post operative records were made of the same parameters as in the study group.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing intestinal anastamosis on an elective or emergency basis

Exclusion Criteria:

* Re laparotomies
* Patients who are immunosuppressed
* Patients with renal failure
* Patients with spinal injuries
* Patients requiring critical care
* Pediatric patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To be able to tolerate early enteral feed | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Kapoor, MS, Study Chair — CMC Hospital; Prerna Gupta, MS, Principal Investigator — CMC Hospital
Locations (1):
- Christian Medical College and Hospital, Ludhiana, Punjab, India